CLINICAL TRIAL: NCT06145399
Title: [18F]-Fluoro-2-Deoxy-D-Glucose and -[18F] Dihydro-Testosterone PET Imaging In Patients Advanced Breast Cancer
Brief Title: A Study of 1 8F-FDHT PET/MRIScans in Women With Breast Cancer
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No accruals
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-299
Record Dates: First submitted 2023-11-16; First posted 2023-11-24 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer; Breast Carcinoma; Metastatic Breast Cancer; Metastatic Breast Carcinoma; Female Breast Cancer
Keywords: Breast Cancer; Breast Carcinoma; Metastatic Breast Cancer; Metastatic Breast Carcinoma; AR+ breast cancer; Progressive metastatic breast cancer; 21-299; Memorial Sloan Kettering Cancer Center; Female Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with Breast Cancer (Experimental): Participants with histologically confirmed AR+ breast cancer
  Interventions: Diagnostic Test: 18F-FDG PET/CT; Diagnostic Test: [18F]-Fluoro-2-Deoxy-D-Glucose and -[18F] Dihydro-Testosterone PET Imaging; Drug: 18F-FDHT

INTERVENTIONS:
Diagnostic Test: 18F-FDG PET/CT — Standard-of-care 18F-FDG PET/CT will be performed using one of the commercially available GE PET/CT scanners
Diagnostic Test: [18F]-Fluoro-2-Deoxy-D-Glucose and -[18F] Dihydro-Testosterone PET Imaging — 18F- FDHT PET/MRI examinations will be performed to evaluate the association between 18F-FDHT uptake and AR expression levels as determined by immunohistochemistry (IHC) in selected lesions.
  Other Names: 18F- FDHT PET/MRI examinations
Drug: 18F-FDHT — 18F- FDHT PET/MRI examinations will be performed to evaluate the association between 18F-FDHT uptake and AR expression levels as determined by immunohistochemistry (IHC) in selected lesions.
  Other Names: [18F]-Fluoro-2-Deoxy-D-Glucose and -[18F] Dihydro-Testosterone

SUMMARY:
The purpose of this study is to see whether 18F-FDHT PET/MRI scans are an effective way of identifying AR-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ECOG performance score of 0-2
* Signed informed consent
* Histologically confirmed AR+ breast cancer

  * All participants under consideration for enrollment will have their tumor specimen tested centrally at MSK; nuclear AR staining ≥ 1% will be considered positive.
* Progressive metastatic breast cancer manifested as increase in evaluable disease OR the appearance of new sites of disease since the date of the last imaging study performed and under consideration for AR-targeted therapy
* Planning to undergo treatment with agents targeting the antiandrogen signaling pathway on a clinical trial

Exclusion Criteria:

* Life expectancy < 3 months
* Pregnancy or lactation
* Participants who cannot undergo scanning because of

  * weight limits
  * devices or implants that are not MRI safe
  * allergies to contrast materials
* CNS only disease on recent imaging

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All participants recruited to the protocol will be women, as breast cancer is primarily a disease of women
Enrollment: 0 (Actual)
Dates: Start 2023-10-24 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Number of lesions that correlate 18F-FDHT uptake with IHC expression of AR | 8 weeks post treatment
  The primary objective is to correlate 18F-FDHT uptake with IHC expression of AR as in selected lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Maxine Jochelson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org